CLINICAL TRIAL: NCT07169929
Title: The Reliability of Measuring Transverse Thalamic Diameter in Determining the Gestational Age as a Fetal Growth Parameter Using 2D Ultrasound
Brief Title: Fetal Transverse Thalamic Diameter and Assessment of Gestational Age as a Fetal Growth Parameter Using 2D Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Assistant professor of Obstetrics and Gynecology, Cairo University
Other Study IDs: Transverse thalamic diameter
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Fetal Conditions
Keywords: Transverse thalamic diameter - fetal growth - 2Dultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy pregnant women who will meet the inclusion criteria and attend the feto-maternal unit
  Interventions: Other: Measurement of fetal transverse thalamic diameter by 2dimensional abdominal ultrasound

INTERVENTIONS:
Other: Measurement of fetal transverse thalamic diameter by 2dimensional abdominal ultrasound — All pregnant women attending the feto-maternal unit with gestational age from 18 weeks to 36 weeks in the obstetrics and gynecology department in the faculty of medicine Cairo university Using curvilinear 2D transabdominal ultrasound probe of ultrasound machine either Voluson E10 GE or Nuewa I9 Elite Mindray.
  The investigators will take all the biometry (Biparietal diameter, head circumference, abdominal circumference, femur length and trans-cerebellar diameter) and exclude any congenital anomalies in the scan.
  Transverse thalamic diameter is to be measured by 2D ultrasound at the standard axial trans-cerebellar plane. A guitar shape representative structure is presented to demarcate the thalamic diameter.
  Calculate the gestational age using transverse thalamic diameter from this equation Transverse thalamic Diameter( in mm)=0.912 x Gestational age in weeks -1.134) ( Sridar P, et al 2020)

SUMMARY:
The thalamus is a nuclear complex which located in the diencephalon of the brain. Its main function is to relay messages which affect the sensory and motor functions in the body. A lot of behavioral functions are accredited to it such as memory, learning, attention and language. (Sridar P,et al 2020) There is an automatic thalamic diameter measurement to estimate the thalamic diameter, with the measurement accuracy as good as the clinical assessment.( Sridar P,et al 2016) Transverse thalamic diameter increased significantly with increasing gestational age, head circumference, and trans-cerebellar diameter linearly, and normal range thalamic charts are presented. The guitar shape provided good reproducibility of thalamic diameter measures. (Sridar P,et al 2020) Also the evaluation of echogenic thalamus is beneficial, and can be considered as a new marker of fetal lung maturity. ( Rasheed FA, et al 2012).

Maternal hyperglycemia was significantly associated with an increase in the widths of fetal posterior lateral ventricles, cavum septum pellucidi, and cisterna magna and a decrease in fetal trans-cerebellar diameter with no difference was found between three groups in terms of fetal thalamus size (Ekin A. et al 2023).

However, little is known about the growth pattern of thalami during fetal life, and virtually nothing is known about the possible association of deviations from the normal growth pattern with the abnormal conditions. There is a study published on fetal thalami which compare the volumes of cerebral structures, including thalami, between two group's normally growing and growth-restricted fetuses and reported lack of significant difference in thalamic volumes between the two groups. (Elshal RS.etal 2023).

During fetal life, the thalamus increases in size between the ages of 20 to 43 weeks of gestation (Tutunji R et al 2018 ) The development of the thalamus is not a unified progress as it shows remarkable dynamism and heterogeneity ( Zheng et al., 2023) For example, before 35 weeks post-menstrual age ,morphological changes were relatively uniform across the thalamus, and after 35 weeks post menstrual age, deformation was more obvious at the rim than in the central part of the thalamus (Liu et al., 2021).

Prospective research ensures focused attention to the structures to be measured, with more clearly imaged by the operator and using variable contrast resolution to ensuring clarity of the measured structure and prevent any artefacts which prevent visualization. .( Sridar P etal 2020) While Ultrasound allows the measurement of the fetal brain in real time and has fewer artefacts from the movement of the fetus, it is operator dependent. (Bookstein S etal 2024).

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with singleton pregnancy with gestational age between 18 to 36 weeks

Exclusion Criteria:

* Women who are not sure of dates and don't have an US report with CRL measured in the first trimester
* Maternal obesity (BMI>35) as abdominal fat cause restriction in taking measurement
* Known case of DM or Hypertension or SLE
* Any fetal head or CNS anomalies
* Any maternal opiates and CNS drugs (methadone) IUGR
* Twins or multiple pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant women who will meet the inclusion criteria and attend the feto-maternal unit in the department of obstetrics and gynecology faculty of medicine Cairo university consent to participate in the research study
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Realibity of transverse thalamic diameter as a parameter for fetal growth | 6months
  Correlation of measuring the transverse thalamic diameter in determining the gestational age between 18 weeks and 36 weeks according to this equation (Transverse thalamic Diameter( in mm)=0.912 x Gestational age in weeks -1.134) ( Sridar P, et al 2020)